CLINICAL TRIAL: NCT03906747
Title: End-of-Life Management Protocol Offered Within Emergency Room: a Multicentre Study (EMPOWER)
Acronym: EMPOWER
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Singapore Clinical Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: HSRG-EoL17Jun001
Record Dates: First submitted 2019-02-25; First posted 2019-04-08 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-03

CONDITIONS: Palliative Care; Emergency Department; Cost Effectiveness
MeSH Terms: conditions — Emergencies | interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients: Patients at their end-of-life (EOL) phase attending the emergency department
  Interventions: Other: Review of medical records
- Family members and next-of-kin of (EOL) patients: Family members and next-of-kin of EOL patients in the emergency department
  Interventions: Other: Interviews, questionnaire and focused group discussions
- Healthcare workers: Comprised of doctors in the emergency department, nurses and general practitioners
  Interventions: Other: Interviews, questionnaire and focused group discussions

INTERVENTIONS:
Other: Interviews, questionnaire and focused group discussions — To determine the effectiveness of the quality of care as perceived by relatives, we will perform a survey during the ED stay, with the next-of-kin to patients who was on the EOL pathway using a questionnaire developed for ED settings. The questionnaire will be administered by the research assistant face-to-face in the emergency department to assess the quality of care and the level of support provided to patients and their families in the last days of life.
  We will also determine the level of staff's knowledge and perception of the EOL care using a locally-designed self-administered anonymous survey.
  A focus group discussion (FGD) will be formed in each hospital to identify the gaps to the current EOL care by structured questionnaire. The group will also make recommendations to improve the quality of the EOL care. There will be separate FGD for: (i) healthcare professionals (ii) family members and (iii) general practitioners who will care for the patient if terminally discharged.
  Groups: Family members and next-of-kin of (EOL) patients; Healthcare workers
Other: Review of medical records — Electronic medical records will be reviewed to collect the following data:
  1. Proportion of patients who fits criteria of EOL who died within 48 hours;
  2. Proportion of patients on EOL pathway who have documentation that patient and/or family are given opportunities to discuss an individualised care plan;
  3. Proportion of patients on EOL pathway who have documentation of an individualised care plan that is followed;
  4. Proportion of patients on EOL pathway who have symptoms who are prescribed with medicines with individualised indications for use, dosage and route of administration
  Groups: Patients

SUMMARY:
End-of-life (EOL) care has garnered increasing recognition and acceptance in the field of emergency medicine. Some emergency departments (EDs) in Singapore have instituted or plan to institute EOL care as part of the workflow. However, the EOL protocols are not standardised across all these EDs. The adherence to and quality of EOL care have not been formally measured in all institutions. Hence, gaps to improve the quality of care have yet to be determined.

The aims are to systematically measure the current quality of EOL care in three Singapore hospital EDs and identify the quality gaps; formulate interventions to address these gaps and implement the improved EOL care; and measure the improvement post-implementation. The investigators hypothesise that the current quality of EOL care in three EDs is suboptimal and the interventions planned will improve the quality of care provided.

The study team plans to conduct an interrupted time series study to detect whether the interventions have an effect significantly greater than any underlying trend over time. The quality of care indicators to be measured are timely identification of patients who require EOL care, adequacy of symptom control based on compliance to prescriptions, opportunities to discuss and develop an individualised care plan, perceived quality of care by healthcare providers and next-of-kin, and cost effectiveness. Planned interventions include refining the protocol with collaboration of content experts in palliative care, education and training of healthcare providers, and addressing specific gaps identified to improve cost effectiveness. The results of this study will form the standardisation and foundation for establishing the national benchmark for quality of EOL care in Singapore EDs.

ELIGIBILITY:
Inclusion Criteria:

* Actively dying patient or high likelihood of mortality within 48 hours
* Family accepts that the goals of care are provision of comfort, symptom relief and respect of dignity
* Patient is not a candidate for cardiopulmonary resuscitation, endotracheal intubation or transfer to the intensive care unit
* Family members want to stay by patient's bedside
* Any of the life-limiting conditions such as chronic frailty with poor functional state and limited reversibility (Karnofski Performance Scale <40%), chronic severe illness with poor prognosis, or other deteriorating conditions and at risk of dying with complications that are not reversible, as subject to the treating clinician's judgment

Exclusion Criteria:

* Vulnerable population e.g. prisoners, pregnant women
* Patients, relatives or staff who refused to participate
* Patients who have been recruited, or had declined participation, in the previous ED attendance(s)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending the emergency department at their end-of-life phase, relatives of such patients and healthcare workers involved with care
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2019-01-18 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality rate within 48 hours of hospital admission | 26 months
  Proportion of patients who fits criteria of EOL who died within 48 hours (patient centred)
Satisfaction assessed by Care of the Dying Evaluation (CODE) questionnaire | 26 months
  Proportion of next-of-kin who perceived that they were adequately supported (family centred)
Satisfaction of healthcare workers with care rendered assessed by a staff survey | 26 months
  Level of satisfaction of with the overall quality of end of life care provision by doctors at ED

SECONDARY OUTCOMES:
Proportion of patients in EOL pathway who have documentation of an individualised care plan, and symptoms who are prescribed with appropriate medicine | 26 months
  Proportion of patients in EOL pathway who have documentation of an individualised care plan, and symptoms who are prescribed with appropriate medicine

CONTACTS AND LOCATIONS:
Locations (3):
- Singapore (3):
  - National University Hospital, Singapore
  - Changi General Hospital, Singapore
  - Khoo Teck Puat Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chua MT, Sen Kuan W, Zheng CQ, Tiah L, Kumar R, Wong YKY, Lin J, Liang S, Mayland CR, Shi L, Ibrahim I, Pal RY. Validation of "Care of the Dying Evaluation" in Emergency Medicine (CODE-EM): pilot phase of end-of-life management protocol offered within emergency room (EMPOWER) study. Ann Palliat Med. 2021 Jun;10(6):6145-6155. doi: 10.21037/apm-21-380. Epub 2021 May 25. PMID 34118856
- [Derived] Yash Pal R, Kuan WS, Tiah L, Kumar R, Wong YKY, Shi L, Zheng CQ, Lin J, Liang S, Segara UC, Yong WC, Chan NGC, Chua MT, Ibrahim I. End-of-life management protocol offered within emergency room (EMPOWER): study protocol for a multicentre study. BMJ Open. 2020 Apr 28;10(4):e036598. doi: 10.1136/bmjopen-2019-036598. PMID 32350018